CLINICAL TRIAL: NCT00342823
Title: Immunogenetics of Visceral Leishmaniasis
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904024; 04-HG-N024
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-06-30

CONDITIONS: Visceral Leishmaniasis
Keywords: Linkage Analysis; Canidate Gene Analysis; Genome Scan; L. Chagasi; Visceral Leishmania
MeSH Terms: conditions — Leishmaniasis, Visceral

SUMMARY:
Visceral leishmaniasis is a potentially fatal disease caused in South America by the protozoan Leishmania chagasi. In neighborhoods with high exposure rates, the outcome of human infection with L. chagasi ranges from asymptomatic to a disseminated wasting disease called visceral leishmaniasis (VL). Several studies document familial clustering of VL in populations at risk. Segregation analyses favor a genetic over an environmental model for susceptibility to L. chagasi infection. A peri-urban outbreak of VL near the Universidade Federal do Rio Grande do Norte (UFRN) in Natal, northeast Brazil, has allowed us to identify endemic neighborhoods with ongoing transmission of L. chagasi infection. Natal is ideal for this study because endemic neighborhoods are easily accessible, people are motivated to cooperate with measures to control VL, and other forms of leishmaniasis are not transmitted in the region. Dr. Jeronimo of the UFRN, and Dr. Mary Wilson at University of Iowa have collected clinical data and DNA from 400 VL families living in these endemic neighborhoods. We have created an unprecedented cohort through which we can identify four distinct phenotypic responses after L. chagasi exposure. We documented familial clustering of L. chagasi infection, and results of both correlation and segregation analyses are consistent with the hypothesis that genetic factors predispose, in part, to the diverse clinical outcomes after infection. Polymorphism in the TNF locus is associated with developing symptomatic as opposed to asymptomatic disease after infection. We recently completed a genome-wide scan of the quantitative immune response (DTH) and identified potential linkage regions on chromosomes 2, 13, 15 and 19. We have also identified a small linkage peak on chromosome 9 for VL. In our ongoing study, we will next perform fine mapping of these regions using dense SNPs to identify genes that may determine susceptibility to L. chagasi infection. Additionally, we will also analyze candidate genes for association/linkage with susceptibility to or protection from L. chagasi disease. We recently identified an association on chromosome 5 with the DTH immune response among two linkage disequilibrium blocks spanning multiple immune related genes.

DETAILED DESCRIPTION:
Visceral leishmaniasis is a potentially fatal disease caused in South America by the protozoan Leishmania chagasi. In neighborhoods with high exposure rates, the outcome of human infection with L. chagasi ranges from asymptomatic to a disseminated wasting disease called visceral leishmaniasis (VL). Several studies document familial clustering of VL in populations at risk. Segregation analyses favor a genetic over an environmental model for susceptibility to L. chagasi infection. A peri-urban outbreak of VL near the Universidade Federal do Rio Grande do Norte (UFRN) in Natal, northeast Brazil, has allowed us to identify endemic neighborhoods with ongoing transmission of L. chagasi infection. Natal is ideal for this study because endemic neighborhoods are easily accessible, people are motivated to cooperate with measures to control VL, and other forms of leishmaniasis are not transmitted in the region. Dr. Jeronimo of the UFRN, and Dr. Mary Wilson at University of Iowa have collected clinical data and DNA from 400 VL families living in these endemic neighborhoods. We have created an unprecedented cohort through which we can identify four distinct phenotypic responses after L. chagasi exposure. We documented familial clustering of L. chagasi infection, and results of both correlation and segregation analyses are consistent with the hypothesis that genetic factors predispose, in part, to the diverse clinical outcomes after infection. Polymorphism in the TNF locus is associated with developing symptomatic as opposed to asymptomatic disease after infection. We recently completed a genome-wide scan of the quantitative immune response (DTH) and identified potential linkage regions on chromosomes 2, 13, 15 and 19. We have also identified a small linkage peak on chromosome 9 for VL. In our ongoing study, we will next perform fine mapping of these regions using dense SNPs to identify genes that may determine susceptibility to L. chagasi infection. Additionally, we will also analyze candidate genes for association/linkage with susceptibility to or protection from L. chagasi disease. We recently identified an association on chromosome 5 with the DTH immune response among two linkage disequilibrium blocks spanning multiple immune related genes.

ELIGIBILITY:
* INCLUSION CRITERIA:

We used three approaches to identify families in endemic neighborhoods, yielding three populations of families.

Population I: A neighborhood to the northeast of the city was identified through a family with two cases of disease.

Population 2: Individuals with suspected VL are admitted to one of three public hospitals in Natal. Families were interviewed and examined if they wished to participate.

Population 3: The neighboring families living closest to population 2 families were identified.

EXCLUSION CRITERIA

Individuals with ongoing illnesses other than VL were excluded from analyses.

Any medical conditions found or suspected based upon history, exam or blood tests were either treated by the investigators or referred to the appropriate medical facility in Natal.

Pregnant women and children less than 1 year were not given any skin test.

No exclusions based on ethnicity were done.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2003-10-20; Study Completion 2010-06-30

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Norte, Natal, Brazil

REFERENCES:
- [Background] Desjeux P. Leishmaniasis. Public health aspects and control. Clin Dermatol. 1996 Sep-Oct;14(5):417-23. doi: 10.1016/0738-081x(96)00057-0. No abstract available. PMID 8889319
- [Background] Wolday D, Berhe N, Akuffo H, Britton S. Leishmania-HIV interaction: immunopathogenic mechanisms. Parasitol Today. 1999 May;15(5):182-7. doi: 10.1016/s0169-4758(99)01431-3. PMID 10322351
- [Background] de Gorgolas M, Miles MA. Visceral leishmaniasis and AIDS. Nature. 1994 Dec 22-29;372(6508):734. doi: 10.1038/372734b0. No abstract available. PMID 7997260